CLINICAL TRIAL: NCT04573335
Title: Health-related Outcomes and Behaviour Changes in a Cohort of Diabetic Population During COVID-19 Pandemic: Results of a Telephonic Survey
Brief Title: Diabetes Outcomes in COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Dr. Saira Burney, Doctor, Services Institute of Medical Sciences, Pakistan
Other Study IDs: 16102019
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Diabetes; Covid19; Isolation, Social
Keywords: COVID-19; diabetes mellitus; telesurvey
MeSH Terms: conditions — Diabetes Mellitus; COVID-19; Social Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes management and follow-up has become a challenge during the COVID-19 pandemic. Nation-wide lockdowns and social distancing measures adopted in an attempt to break the chain of COVID-19 transmission have significantly disrupted routine care and follow-up of diabetes. In the health sector, especially in low-income countries such as Pakistan, there has been a shift of resources and staff reassignment from stable chronic illnesses to support COVID-19 pandemic. Disruption of routine outpatient health services and travel restrictions increase the risk of worsening diabetes control and diabetes-related health outcomes. Additionally, social isolation amidst an atmosphere of fear and uncertainty contributes to stress further affecting glycaemic control.

DETAILED DESCRIPTION:
An observational cross-sectional study was conducted using telephone interview method in Diabetes Management Centre (DMC), Services hospital, Lahore. The study participants were 1282 diabetic patients selected randomly from electronic medical record (EMR) database of the Centre. A structured questionnaire was used to evaluate parameters which included patients' demographic information; diabetes self-care and general health profile; COVID-related questions and its impact on quality of life (QoL); financial and social support issues.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and type 2 diabetic patients registered with Diabetes Management Centre, Services hospital, Lahore, Pakistan.

Exclusion Criteria:

* Patients lacking telephonic contact or with invalid contact numbers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic subjects already registered with and on regular follow-up with DMC and had visited DMC for consultation more than once between 1st August 2019 to 15th March 2020.
Sampling Method: Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | during 3months of lockdown
  Death due to diabetes-related complications or otherwise

SECONDARY OUTCOMES:
COVID-19 illness | During 3months of lockdown
  %age of participants with one or more symptoms of fever, sore throat, cough, dyspnoea

CONTACTS AND LOCATIONS:
Overall Officials: Saira Burney, MB;FRCP (Edin), Principal Investigator — SIMS
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No